CLINICAL TRIAL: NCT00460278
Title: A Phase 1 Dose-Escalation Study of the Safety and Pharmacokinetics of XL418 Administered Orally Daily to Subjects With Solid Tumors
Brief Title: Study of XL418 in Adults With Solid Tumors
Status: Suspended | Phase: Phase 1 | Type: Interventional
Why Stopped: Enrollment suspended due to low drug exposure.
Sponsor: Exelixis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XL418-001
Record Dates: First submitted 2007-04-11; First posted 2007-04-13 (Estimated); Last update posted 2008-06-04 (Estimated); Status verified 2008-06

CONDITIONS: Cancer; Solid Tumors
Keywords: Cancer; Solid Tumors
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: XL418

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of XL418 in subjects with solid tumors. XL418 is a new chemical entity that inhibits a spectrum of targets, including Akt and p70S6K, that mediate PI3 Kinase / PTEN signaling.

ELIGIBILITY:
Inclusion Criteria:

1. The subject has a histologically confirmed solid tumor that is metastatic or unresectable, for which standard curative or palliative measures do not exist or are no longer effective, and there are no known therapies to prolong survival.
2. The subject has disease that is assessable by tumor marker, physical, or radiologic means.
3. The subject is ≥18 years old.
4. The subject's weight is ≥55 kg and ≤120 kg.
5. The subject has an ECOG (Eastern Cooperative Oncology Group) performance status ≤2.
6. The subject has adequate organ and marrow function.
7. For subjects who are to be enrolled into the expanded MTD cohort:

   1. tumor tissue amenable to serial biopsy; and
   2. additional informed consent.
8. The subject is capable of understanding the protocol and has signed the informed consent document.
9. Sexually active subjects (male and female) must use medically acceptable methods of contraception during the course of the study.
10. Female subjects of childbearing potential must have a negative serum pregnancy test at screening.
11. The subject has a normal fasting blood glucose level at screening.
12. If a subject has received more than three prior regimens of cytotoxic chemotherapy, more than two biological regimens, or more than 3000 cGy to areas containing substantial marrow, the principal investigator (PI) and the sponsor will discuss subject suitability prior to enrollment.
13. The subject has had no other diagnosis of malignancy (unless non-melanoma skin cancer, in situ carcinoma of the cervix, or a malignancy diagnosed ≥5 years ago, with no evidence of disease for 5 years prior to screening for this study).

Exclusion Criteria:

1. The subject has received anticancer treatment (eg, chemotherapy, radiotherapy, cytokines, or hormones) within 30 days (6 weeks for nitrosoureas or mitomycin C) before the first dose of study drug.
2. The subject has received radiation to ≥25% of his or her bone marrow within 30 days of treatment with XL418.
3. The subject has not recovered either to Grade ≤1 from adverse events (AEs) or to within 10% of baseline values due to investigational or other agents administered more than 30 days prior to study enrollment.
4. The subject has received another investigational agent within 30 days of the first dose of study drug.
5. The subject has known brain metastases.
6. The subject is known to have diabetes.
7. The subject has an uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, hypertension, symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia.
8. The subject has psychiatric illness/social situations that would limit compliance with study requirements.
9. The subject is pregnant or breast feeding.
10. The subject is known to be positive for the human immunodeficiency virus (HIV).
11. The subject has a known allergy or hypersensitivity to any of the components of the XL418 formulation.
12. The subject has a baseline QTc interval >450 ms.
13. The subject is unwilling or unable to abide by the study protocol or cooperate fully with the investigator or designee.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2007-04

PRIMARY OUTCOMES:
Safety, tolerability, and maximum tolerated dose of XL418 with daily oral administration

SECONDARY OUTCOMES:
Plasma pharmacokinetics and pharmacodynamic effects of daily oral administration of XL418

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Wayne State University, Detroit, Michigan
  - South Texas Accelerated Research Therapeutics, San Antonio, Texas